CLINICAL TRIAL: NCT04220853
Title: Changes in Nasal Airflow Parameters After Septoplasty and Turbinoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-Nasal_obstruction
Record Dates: First submitted 2019-09-04; First posted 2020-01-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Nasal Obstruction; Nasal Septum; Deviation; Nasal Mucosa Hypertrophy
Keywords: nasal obstruction; septoplasty; turbinoplasty; nasal mucosa; nasal septum
MeSH Terms: conditions — Nasal Obstruction | interventions — Rhinomanometry; Rhinometry, Acoustic

STUDY DESIGN:
Intervention Model Description: The patients will be divided into three parallel groups, depending on the indicated surgery - septoplasty, turbinoplasty, and septoplasty plus turbinoplasty.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Septoplasty (Experimental): The patients indicated for septoplasty will be included in this arm. The patients will undergo rhinomanometry and acoustic rhinometry after the surgery.
  Interventions: Diagnostic Test: Rhinomanometry in patients after septoplasty and/or turbinoplasty; Diagnostic Test: Acoustic rhinometry in patients after septoplasty and/or turbinoplasty
- Turbinoplasty (Experimental): The patients indicated for turbinoplasty will be included in this arm. The patients will undergo rhinomanometry and acoustic rhinometry after the surgery.
  Interventions: Diagnostic Test: Rhinomanometry in patients after septoplasty and/or turbinoplasty; Diagnostic Test: Acoustic rhinometry in patients after septoplasty and/or turbinoplasty
- Septoplasty and turbinoplasty (Experimental): The patients indicated for septoplasty and turbinoplasty will be included in this arm. The patients will undergo rhinomanometry and acoustic rhinometry after the surgery.
  Interventions: Diagnostic Test: Rhinomanometry in patients after septoplasty and/or turbinoplasty; Diagnostic Test: Acoustic rhinometry in patients after septoplasty and/or turbinoplasty

INTERVENTIONS:
Diagnostic Test: Rhinomanometry in patients after septoplasty and/or turbinoplasty — Rhinomanometry is an examination used to assess changes in resistance and airflow in patients after septoplasty and/or turbinoplasty.
Diagnostic Test: Acoustic rhinometry in patients after septoplasty and/or turbinoplasty — Acoustic rhinometry is an examination used to assess changes in the cross-sectional area of the nasal passage in patients after septoplasty and/or turbinoplasty.

SUMMARY:
Pathological-anatomical changes in the nasal cavity (nasal septum/perforation, mucosal hypertrophy) negatively affect nasal airflow, increase resistance - cause nasal obstruction and are often an indication for surgery.

The aim of the study is to examine nasal airflow parameters after septoplasty and turbinoplasty .

DETAILED DESCRIPTION:
Pathological-anatomical changes in the nasal cavity (nasal septum/perforation, mucosal hypertrophy) negatively affect nasal airflow, increase resistance - cause nasal obstruction and are often an indication for surgery.

The aim of the study is to examine nasal airflow parameters at pre-defined intervals in patients after septoplasty and turbinoplasty .

ELIGIBILITY:
Inclusion Criteria:

* patients with nasal obstruction (nasal septal deviation, hypertrophy of nasal mucosa)
* 18 to 70 Years
* patient capable of general anesthesia
* signing of the informed consent

Exclusion Criteria:

- patient incapable of general anesthesia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in resistance | 6 and 12 weeks after surgery
  Changes in resistance (measured in Pa-s/ml - Pascal-second/millilitre) will be assessed with rhinomanometry 6 and 12 weeks after surgery.
Changes in airflow | 6 and 12 weeks after surgery
  Changes in airflow (measured in ml/s - millilitres/second) will be assessed with rhinomanometry 6 and 12 weeks after surgery.
Changes in the cross-sectional area of the nasal passage | 6 and 12 weeks after surgery
  Changes in the cross-sectional area of the nasal passage will be assessed with acoustic rhinometry 6 and 12 weeks after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marek Plášek, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Parthasarathi K, Christensen JM, Alvarado R, Barham HP, Sacks R, Harvey RJ. Airflow and symptom outcomes between allergic and non-allergic rhinitis patients from turbinoplasty. Rhinology. 2017 Dec 1;55(4):332-338. doi: 10.4193/Rhin16.210. PMID 28888024
- [Background] Ottaviano G, Fokkens WJ. Measurements of nasal airflow and patency: a critical review with emphasis on the use of peak nasal inspiratory flow in daily practice. Allergy. 2016 Feb;71(2):162-74. doi: 10.1111/all.12778. PMID 26447365
- [Background] Borojeni AAT, Garcia GJM, Moghaddam MG, Frank-Ito DO, Kimbell JS, Laud PW, Koenig LJ, Rhee JS. Normative ranges of nasal airflow variables in healthy adults. Int J Comput Assist Radiol Surg. 2020 Jan;15(1):87-98. doi: 10.1007/s11548-019-02023-y. Epub 2019 Jul 2. PMID 31267334
- [Background] Mlynski G, Grutzenmacher S, Plontke S, Mlynski B, Lang C. Correlation of nasal morphology and respiratory function. Rhinology. 2001 Dec;39(4):197-201. PMID 11826688